CLINICAL TRIAL: NCT00929994
Title: Effects of Cardiac Rehabilitation for Individuals With Transient Ischemic Attack
Status: Completed | Type: Observational
Sponsor: Toronto Rehabilitation Institute (Other)
Collaborators: Heart and Stroke Foundation of Canada (Other)
Responsible Party: Principal Investigator, Dina Brooks, Professor, Toronto Rehabilitation Institute
Other Study IDs: Brooks - 001
Record Dates: First submitted 2009-06-29; First posted 2009-06-30 (Estimated); Results first posted 2019-04-23 (Actual); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Transient Ischemic Attack
Keywords: cardiac rehab
MeSH Terms: conditions — Ischemic Attack, Transient | interventions — Cardiac Rehabilitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Exercise: Following a 3 month non intervention period, participants will participate in Cardiac Rehabilitation, carrying out an exercise program which will last 6 months and combine both resistance and aerobic training.
  Interventions: Behavioral: Cardiac Rehabilitation

INTERVENTIONS:
Behavioral: Cardiac Rehabilitation — Individualized cardiac rehabilitation for 6 months, including health education sessions, as well as supervised exercise classes which include aerobic and resistance training.

SUMMARY:
It is hypothesized that the addition of formal cardiac rehabilitation to standard care will result in long-term improvements in cardiovascular fitness and functional capacity in individuals who have suffered a transient ischemic attack (TIA) or minor stroke.

Furthermore, it is proposed that the addition of cardiac rehabilitation will influence depressive symptoms and cognition.

DETAILED DESCRIPTION:
A transient ischemic attack (TIA) is defined as an episode of neurological dysfunction caused by focal brain ischemia lasting less than 24 hours. Once an individual has suffered a TIA, preventative measures can be taken to target modifiable risk factors, one of which is physical inactivity. The current proposal focuses on the use of an established model of care (cardiac rehabilitation (CR)) and applies it to those who have suffered a TIA in order to maximize physical activity and minimize risk of future cardiovascular events. This will be a one-group pre/post design study with a 3 month non-intervention period. Participants will undergo measures at baseline and 3 months (non intervention period) then after 6 months of cardiac rehabilitation (cardiovascular fitness, 6 minute walk test, cognition, and depressive symptoms).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with TIA
* Three months post-TIA
* Ability to understand the process and instructions for exercise training and provide informed consent

Exclusion Criteria:

* Resting Blood Pressure greater than 160/100 despite medication
* Other cardiovascular morbidity which would limit exercise tolerance (heart failure, abnormal BP responses or STsegment depression > 2 mm, symptomatic aortic stenosis, complex arrhythmias)
* Current and extensive exercise participation
* Hypertrophic Cardiomyopathy
* Unstable Angina
* Orthostatic BP decrease of > 20 mm Hg with symptoms
* Other musculoskeletal impairments which would limit the participants ability to walk sufficient durations
* Pain or other co-morbidities (e.g., unclipped aneurysms, uncontrolled seizures etc.) which would preclude participation
* Cognitive or behavioural issues that would limit participation in exercise testing and training

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: TIA
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2010-03; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dina Brooks, PhD, Principal Investigator — Toronto Rehabilitation Institute; William E McIllroy, PhD, Principal Investigator — University of Waterloo; Paul Oh, MD, Principal Investigator — Toronto Rehabilitation Institute; Sandra Black, MD, Principal Investigator — Sunnybrook and Women's College Health Centre
Locations (1):
- Toronto Rehabilitation Institute - Rumsey Center, Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Exercise: Participants will participate in Cardiac Rehabilitation, carrying out an exercise program which will last 6 months and combine both resistance and aerobic training. There will be a 3 month non-intervention period preceding the exercise program.
  Cardiac Rehabilitation: Individualized cardiac rehabilitation for 6 months, including health education sessions, as well as supervised exercise classes which include aerobic and resistance training.
Period: Overall Study
Arm/Group | Exercise
Started | 20
Completed | 14
Not Completed | 6
Not completed — Withdrawal by Subject | 1
Not completed — medical issue unrelated to intervention | 4
Not completed — employment | 1

BASELINE CHARACTERISTICS:
Groups:
- Exercise: Participants in this group will participate in Cardiac Rehabilitation, carrying out an exercise program which will last 6 months and combine both resistance and aerobic training.
  Cardiac Rehabilitation: Individualized cardiac rehabilitation for 6 months, including health education sessions, as well as supervised exercise classes which include aerobic and resistance training.
Arm/Group | Exercise
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 7
Region of Enrollment [Number; unit: participants]
  Canada | 20

OUTCOME MEASURES:

1. Primary Outcome: Functional Walk Test
Description: 6 minute walk test: the longest distance a person can walk for a duration of 6 minutes
Time Frame: Baseline, 3 months, 6 months (Six Minute Walk Distance)
Population: Transient Ischemic Attack participants who completed the 6 month intervention.
Measure: Mean (Standard Deviation); unit: meters
Groups:
- Exercise: Participants in this group will participate in Cardiac Rehabilitation, carrying out an exercise program which will last 6 months and combine both resistance and aerobic training. A 3 month non-intervention period will precede the 6 month cardiac rehabilitation training program.
  Cardiac Rehabilitation: Individualized cardiac rehabilitation for 6 months, including health education sessions, as well as supervised exercise classes which include aerobic and resistance training.
Arm/Group | Exercise
Number analyzed (Participants) | 14
meters
  Baseline | 498.4 (95.2)
  3 months | 503.2 (111.1)
  6 months | 564.2 (139.6)
Statistical Analysis 1: Comparison: Exercise; With 1 group and 3 test times, a repeated measures analysis of variance of 6MWD, was utilized between the 3 test times 0, 3, and 6 months). A Bonferroni correction for multiple testing was used for post hoc contrasts; Test type: Other; p = 0.06, ANOVA — A Bonferroni correction for multiple testing was used for post hoc contrasts. Assumption of sphericity was met for all analyses determined by the Mauchley test of sphericity (all >.05)
Statistical Analysis 2: Comparison: Exercise; Test type: Superiority; p = 0.06, t-test, 2 sided

2. Primary Outcome: Cardiovascular Fitness (VO2peak)
Description: To measure cardiovascular fitness, a stress test on either an upright cycle ergometer (Ergoselect 200P, Germany), or a treadmill (same modality pre- and post-training) was performed depending on patient balance and comfort.
Time Frame: Baseline (after the 3 month non-intervention period) and after 6 months of participation.
Measure: Mean (Standard Deviation); unit: ml/kg/min
Arm/Group | Exercise
Number analyzed (Participants) | 14
ml/kg/min
  Baseline | 16.7 (5)
  6 months | 19.1 (4.6)
Statistical Analysis 1: Comparison: Exercise; Test type: Superiority; p = 0.01, t-test, 2 sided

3. Secondary Outcome: Center for Epidemiologic Studies Depression Scale (CES-D).
Description: Depressive symptoms using the validated Center for Epidemiologic Studies Depression Scale (CES-D). This is a score from a 20 item questionnaire with minimum value of 0 and maximum value of 60 with higher numbers indicated greater depressive symptoms (worse).
Time Frame: Baseline and 3 months (non-intervention period), after 6 months of cardiac rehabilitation participation
Population: Transient Ischemic Attack. Two patients did not complete questionnaires.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Exercise: Participants in this group will participate in Cardiac Rehabilitation, carrying out an exercise program after a 12 week period of non intervention which will last 6 months and combine both resistance and aerobic training.
  Cardiac Rehabilitation: Individualized cardiac rehabilitation for 6 months, including health education sessions, as well as supervised exercise classes which include aerobic and resistance training.
Arm/Group | Exercise
Number analyzed (Participants) | 12
score on a scale
  Baseline | 6.5 (6)
  3 months | 7.6 (5)
  6 months | 4.3 (5.2)
Statistical Analysis 1: Comparison: Exercise; With 1 group and 3 test times, a repeated measures analysis of variance with pairwise comparisons of CES-D was utilized between the 3 test times baseline, 3 and 6 months; Test type: Superiority; p = 0.04, ANOVA — A Bonferroni correction for multiple testing was used for post-hoc contrasts

4. Secondary Outcome: Cognition
Description: Montreal Cognitive Assessment. The MoCA score ranges from 0 to 30 points with a higher score indicating better cognitive function.
Time Frame: Baseline and 3 months (non-intervention period), after 6 months of cardiac rehabilitation participation
Population: TIA. Three subjects did not complete the assessment at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Exercise: Following a 3 month non intervention period, participants in this group will participate in Cardiac Rehabilitation, carrying out an exercise program which will last 6 months and combine both resistance and aerobic training.
  Cardiac Rehabilitation: Individualized cardiac rehabilitation for 6 months, including health education sessions, as well as supervised exercise classes which include aerobic and resistance training.
Arm/Group | Exercise
Number analyzed (Participants) | 11
units on a scale
  Baseline | 26.5 (2.4)
  3 months | 26.8 (3.4)
  6 months | 27.1 (2)
Statistical Analysis 1: Comparison: Exercise; With 1 group and 3 test times, a repeated measures analysis of variance with pairwise comparisons of MoCA was utilized between the 3 test times (-3, 0 and 6 months). A Bonferroni correction for multiple testing was used for post-hoc contrasts; Test type: Superiority; p > 0.05, ANOVA — A Bonferroni correction for multiple testing was used for post-hoc contrasts

ADVERSE EVENTS:
Groups:
- Exercise: Participants will participate in Cardiac Rehabilitation, carrying out an exercise program which will last 6 months and combine both resistance and aerobic training. There will be a 3 month non-intervention period preceding cardiac rehabilitation.
  Cardiac Rehabilitation: Individualized cardiac rehabilitation for 6 months, including health education sessions, as well as supervised exercise classes which include aerobic and resistance training.
Arm/Group | Exercise
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

LIMITATIONS AND CAVEATS:
This study was conducted in a single centre located in a large city centre and may lack generalizability to other programs, including those where CR services are not publicly funded.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No